CLINICAL TRIAL: NCT06479837
Title: Modeling Host-Pathogen Interaction Using Lymphoid Organoids
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002062; 002062-I
Record Dates: First submitted 2024-06-27; First posted 2024-06-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-02

CONDITIONS: Staphylococcal Infections
Keywords: Organoid; Staphylococcus; Host-pathogen Interactions
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tonsillectomy Patients: Patients undergoing tonsillectomy as part of their clinical care

SUMMARY:
Background:

Staphylococcus aureus (S.aureus) are bacteria that can make people sick. Sometimes, an S. aureus infection can develop inside the spine; these infections can lead to paralysis and death. Researchers do not know how S. aureus interacts with a person s cells to cause infections in the spine.

Objective:

To learn how S. aureus interacts with cells in the body using tissues from tonsils discarded after standard surgery to remove them.

Eligibility:

People aged 2 years and older who are scheduled to have their tonsils removed.

Design:

Researchers will select participants for the study based on review of their existing medical records, including results of blood tests; any imaging scans, including x-rays; and reports about tissue specimens.

Participants will answer questionnaires about their health and past infections. They can do this online or on paper.

Participants will collect a nasal swab 1 week before their surgery. They will be given a tool that looks like a long cotton swab. They will twirl it around inside their nose. The swab will pick up cells and fluids that will be used for research.

After their surgery, the participant s surgeon will save samples of tonsil tissue. The surgeon will send these tissue samples and the nasal swab to researchers at the NIH.

These tissues and the swab will be used in studies to help researchers understand how S. aureus interacts with cells in the body. They hope these studies will help them find better ways to treat S. aureus infections.

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

The purpose of this study is to collect tonsil tissues that are routinely discarded after tonsillectomy procedures to develop lymphoid organoid models to evaluate host-pathogen interactions in human health and disease. One such interaction is the human immunotolerance mechanism to the Chemotaxis Inhibitory Protein of S. aureus (CHIPS).

OBJECTIVES:

Primary Objectives:

-Develop a lymphoid organoid model from discarded human tonsils and determine and compare the human immunologic signatures of primary exposure, within the "antigenic sin" contexts of re-exposure, and with repeated exposures to CHIPS.

Secondary Objective:

-Modulate anti-CHIPS IgG4 class switching through variation of primary and costimulatory signals.

ENDPOINTS:

Primary Endpoints:

Differences between the following within the "antigenic sin" contexts of re-exposure, and with repeated exposures to CHIPS:

* Immune cell composition.
* Anti-CHIPS antibody levels, including total and subclasses of IgG and their neutralizing capacity.
* Cytokine levels.
* Activation-induced cytidine deaminase (AID) levels.
* Single-cell inference of class switch recombination (sciCSR).

Secondary Endpoints:

Differences between the following modulation of primary and costimulatory signals:

* Immune cell composition.
* Anti-CHIPS antibody levels, including total and subclasses of IgG and their neutralizing capacity.
* Cytokine levels.
* AID levels.
* sciCSR

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

* Aged >=2 yrs.
* Undergoing tonsillectomy as part of their clinical care.
* Able to provide informed consent (for ages >=18 years) or has a parent or guardian who can provide informed consent on their behalf (for ages <18 yrs).
* Willing to allow samples and data to be stored and shared for future secondary research.
* Willing to allow future genetic testing on their biospecimens.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Active infection.
* Active tonsilitis.
* Pregnant.
* Diagnosed with an immunosuppressive condition or currently taking immunosuppressive medications.
* Current or past intravenous drug use.
* Any condition that, in the judgment of the investigator, may put the participant at undue risk or make them unsuitable for participation in the study

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing tonsillectomy as part of their clinical care at hospitals and pediatric ear nose and throat (ENT) practices in the US will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2043-12-01 (Estimated); Study Completion 2044-12-01 (Estimated)

PRIMARY OUTCOMES:
Immune cell composition | At time of collection
  Develop a lymphoid organoid model from discarded human tonsils and determine and compare the human immunologic signatures of primary exposure, within the "antigenic sin" contexts of re-exposure, and with repeated exposures to CHIPS.
Anti-CHIPS antibody levels, including total and subclasses of IgG and their neutralizing capacity | At time of collection
  Develop a lymphoid organoid model from discarded human tonsils and determine and compare the human immunologic signatures of primary exposure, within the "antigenic sin" contexts of re-exposure, and with repeated exposures to CHIPS.
Cytokine levels | At time of collection
  Develop a lymphoid organoid model from discarded human tonsils and determine and compare the human immunologic signatures of primary exposure, within the "antigenic sin" contexts of re-exposure, and with repeated exposures to CHIPS.
Activation-induced cytidine deaminase (AID) levels | At time of collection
  Develop a lymphoid organoid model from discarded human tonsils and determine and compare the human immunologic signatures of primary exposure, within the "antigenic sin" contexts of re-exposure, and with repeated exposures to CHIPS.
Single-cell inference of class switch recombination (sciCSR) | At time of collection
  Develop a lymphoid organoid model from discarded human tonsils and determine and compare the human immunologic signatures of primary exposure, within the "antigenic sin" contexts of re-exposure, and with repeated exposures to CHIPS.

SECONDARY OUTCOMES:
Immune cell composition | At time of collection
  Primary signals such as antigen characteristics, and secondary signals such as cytokines have been implicated in class switching to IgG4 but have not been defined with respect to CHIPS. Varying these signals and evaluating: 1) organoid immune cell composition, 2) antibody and 3) cytokines levels, and indicators of class switching such as 4) AID and 5) sciCSR levels, will enable us to evaluate modulation of human immunotolerance to CHIPS.
Anti-CHIPS antibody levels, including total and subclasses of IgG and their neutralizing capacity | At time of collection
  Primary signals such as antigen characteristics, and secondary signals such as cytokines have been implicated in class switching to IgG4 but have not been defined with respect to CHIPS. Varying these signals and evaluating: 1) organoid immune cell composition, 2) antibody and 3) cytokines levels, and indicators of class switching such as 4) AID and 5) sciCSR levels, will enable us to evaluate modulation of human immunotolerance to CHIPS.
Cytokine levels | At time of collection
  Primary signals such as antigen characteristics, and secondary signals such as cytokines have been implicated in class switching to IgG4 but have not been defined with respect to CHIPS. Varying these signals and evaluating: 1) organoid immune cell composition, 2) antibody and 3) cytokines levels, and indicators of class switching such as 4) AID and 5) sciCSR levels, will enable us to evaluate modulation of human immunotolerance to CHIPS.
Activation-induced cytidine deaminase (AID) levels | At time of collection
  Primary signals such as antigen characteristics, and secondary signals such as cytokines have been implicated in class switching to IgG4 but have not been defined with respect to CHIPS. Varying these signals and evaluating: 1) organoid immune cell composition, 2) antibody and 3) cytokines levels, and indicators of class switching such as 4) AID and 5) sciCSR levels, will enable us to evaluate modulation of human immunotolerance to CHIPS.
Single-cell inference of class switch recombination (sciCSR) | At time of collection
  Primary signals such as antigen characteristics, and secondary signals such as cytokines have been implicated in class switching to IgG4 but have not been defined with respect to CHIPS. Varying these signals and evaluating: 1) organoid immune cell composition, 2) antibody and 3) cytokines levels, and indicators of class switching such as 4) AID and 5) sciCSR levels, will enable us to evaluate modulation of human immunotolerance to CHIPS.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Otto, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No
Experiments will be conducted in groups of 5 to 16 organoids and will be reported according to experimental groups. Participant data will not be reported individually.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002062-I.html